CLINICAL TRIAL: NCT07110259
Title: Application of the Artificial Intelligence-Based Gene Mutation Prediction Tool DeepGEM in Patients With Non-Small Cell Lung Cancer (NSCLC): A Prospective, Multicenter, Randomized Controlled Trial
Brief Title: AI-Based DeepGEM Tool for Predicting Gene Mutations in NSCLC Patients: A Randomized Controlled Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jianxing He (Other)
Collaborators: Guangzhou Kingmed Diagnostics Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Jianxing He, Clinical Professor, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NSCLC-DeepGEM-RCT-2025
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Non Small Cell Lung Caner
Keywords: Artificial intelligence; gene mutations
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DeepGEM-Informed Group (Experimental): Participants whose clinicians are provided with DeepGEM-predicted mutation status (EGFR/ALK/ROS1). Physicians may choose to proceed with molecular testing and initiate targeted therapy based on AI predictions.
  Interventions: Other: DeepGEM-guided Molecular Testing and Treatment
- Standard Care Group (Active Comparator): Participants whose clinicians do not receive DeepGEM prediction results and manage the case per standard diagnostic and treatment protocols without AI support.
  Interventions: Other: Standard Diagnostic Pathway

INTERVENTIONS:
Other: DeepGEM-guided Molecular Testing and Treatment — Artificial intelligence-based mutation prediction using DeepGEM to guide clinical decision-making for molecular testing and therapy selection.
  Arms: DeepGEM-Informed Group
Other: Standard Diagnostic Pathway — DeepGEM is used for eligibility screening, but its results are withheld. Clinicians manage patients per standard diagnostic and treatment practices.
  Arms: Standard Care Group

SUMMARY:
This prospective, multicenter, randomized controlled trial aims to evaluate the clinical utility of DeepGEM, an artificial intelligence (AI)-based mutation prediction tool based on histopathological whole-slide images, in patients with non-small cell lung cancer (NSCLC). The study will assess whether DeepGEM can facilitate molecular testing, increase targeted therapy utilization, and improve survival outcomes in a real-world clinical setting. Patients with stage II-IV treatment-naïve NSCLC and qualified pathology slides for DeepGEM analysis will be enrolled. Eligible participants with AI-predicted EGFR, ALK, or ROS1 mutations will be randomized in a 4:1 ratio to either the DeepGEM-informed group (clinicians can access AI results to guide further testing and treatment) or the standard care group (clinicians are blinded to AI results and follow routine care).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years, inclusive, at the time of enrollment.
* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) with clinical stage II-IV as per the 8th edition of the AJCC staging system.
* Availability of qualified histopathological whole-slide images that can be reviewed through the KindMED system(DeepGEM).
* Successful mutation prediction of EGFR, ALK, or ROS1 by the DeepGEM AI tool.
* No prior systemic anti-cancer therapy, including chemotherapy, targeted therapy, or immunotherapy.
* Willing and able to comply with study requirements, including follow-up and treatment; written informed consent must be provided.

Exclusion Criteria:

* Prior systemic anti-tumor therapy (chemotherapy, radiotherapy, targeted therapy-including but not limited to monoclonal antibodies or tyrosine kinase inhibitors) before enrollment.
* Failure of DeepGEM analysis or unqualified histopathological image quality.
* History of any other malignancy within the past 5 years, except for adequately treated basal cell carcinoma of the skin or in situ carcinoma (e.g., cervical carcinoma in situ).
* Cognitive or psychological barriers to understanding or accepting AI-based prediction or molecular testing.
* Pregnant or breastfeeding women, or women of childbearing potential who are not using effective contraception.
* Any other clinical condition that, in the opinion of the investigators, may interfere with the study protocol or compromise participant safety, including poor compliance with study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 950 (Estimated)
Dates: Start 2025-07-31 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From randomization to death from any cause, assessed up to 36 months
  Comparison of OS between the DeepGEM-informed group and the standard care group.
Targeted Therapy Utilization Rate | Up to 6 months post-randomization
  Proportion of participants receiving molecularly matched targeted therapies based on standard genetic testing.

SECONDARY OUTCOMES:
Molecular Testing Rate | Up to 3 months
  Proportion of participants who undergo molecular testing after initial DeepGEM prediction.
Prediction Concordance | Up to 3 months
  Concordance between DeepGEM-predicted mutation status and results from PCR or NGS molecular testing.
Cost-effectiveness of DeepGEM | Up to 12 months
  Evaluation of cost per targeted therapy initiated and cost per life-year gained in the DeepGEM group versus standard care.

IPD SHARING:
Plan to Share IPD: No